CLINICAL TRIAL: NCT03572439
Title: Identification of the Sensory Level Block to Cold During Epidural Analgesia for Labor: A Cohort Study to Determine the Influence of the Direction of Testing (Anesthetized Area to Non-anesthetized Area Versus Non-anesthetized to Anesthetized Area)
Brief Title: Identification of the Sensory Level Block to Cold During Epidural Analgesia for Labor: A Cohort Study to Determine the Influence of the Direction of Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-05
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Labor Pain
Keywords: epidural; sensory block level; dermatome
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cephalad to caudal (Active Comparator): Sensory block level check using ice, moving from cephalad to caudal
  Interventions: Diagnostic Test: Sensory block level check using ice
- Caudal to cephalad (Active Comparator): Sensory block level check using ice, moving from caudal to cephalad
  Interventions: Diagnostic Test: Sensory block level check using ice

INTERVENTIONS:
Diagnostic Test: Sensory block level check using ice — Patients are asked to report when the ice feels as cold as it does on the forehead.

SUMMARY:
Assessment of the upper sensory block level during neuraxial analgesia for labor and delivery is an essential component of clinical management and patient safety. A variety of methods have been used for testing the sensory block such as cold, light touch, sharp touch or prick and transcutaneous electrical stimulation. In addition to the diversity of methods, the endpoints used by investigators have also been variable, considering total or partial responses as endpoints. Not surprisingly, a variable sensory block level could be identified as a result of the different methods and types of question asked by the examiner. Another complicating factor is the lack of standardization of the direction of the testing as it relates to anesthetized and non-anesthetized areas. This lack of standardization may result in a difference of several dermatomes in the level that two different assessors might record for the same patient. Considering a clinical research scenario, it may be difficult to replicate results and implement clinical practices. The objective of this study is to determine the degree of agreement between two methods of assessing the sensory block level to cold in women receiving epidural analgesia for labor (anesthetized to non-anesthetized segments versus non-anesthetized to anesthetized segments).

ELIGIBILITY:
Inclusion Criteria:

* patients who request and have no contraindications to receive epidural analgesia
* capable of understanding and signing the written informed consent
* have no language barrier to respond to the level of sensory block assessment
* have no conditions that could compromise their sensitivity to cold.

Exclusion Criteria:

* patients who refuse to sign consent
* epidural analgesia is contraindicated

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
The lower sensory block level to cold | 1 hour
  The sensory block level will be defined as: the dermatome at which and below which there is complete loss of sensation to cold
The upper sensory block level to cold | 1 hour
  The sensory block level will be defined as: the dermatome at which and below which there is still partial sensation to cold

SECONDARY OUTCOMES:
Patient satisfaction | 20 minutes
  Patients will be asked to report satisfaction with the test done from 0-10 (0=very uncomfortable 10=most comfortable
The lower sensory block level to cold | 2 hours
  The sensory block level will be defined as: the dermatome at which and below which there is complete loss of sensation to cold
The upper sensory block level to cold | 2 hours
  The sensory block level will be defined as: the dermatome at which and below which there is still partial sensation to cold

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Souza Soares EC, Balki M, Downey K, Ye XY, Carvalho JCA. Assessment of sensory block during labour epidural analgesia: a prospective cohort study to determine the influence of the direction of testing. Can J Anaesth. 2022 Jun;69(6):750-755. doi: 10.1007/s12630-022-02228-x. Epub 2022 Mar 14. PMID 35289377